CLINICAL TRIAL: NCT01177657
Title: Case-control Study to Evaluate the Vaccine Effectiveness of Rotarix™ Against Rotavirus Severe Gastroenteritis (RV SGE) Among Hospitalized Children Born After 6 March 2006 and at Least 12 Weeks of Age, in Belem, Brazil
Brief Title: Study to Evaluate the Effectiveness of Rotarix™ Against Severe Gastroenteritis Among Hospitalized Children in Brazil
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111562
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Rotavirus Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample

GROUPS / COHORTS (3):
- Gastroenteritis cohort: Children born after 6 March 2006, at least 12 weeks of age and hospitalized for rotavirus severe gastroenteritis
  Interventions: Procedure: Stool sampling
- Hospital control cohort: Children hospitalized for non gastroenteritis causes
- Neighbourhood control cohort: Children without any symptoms of gastroenteritis or severe gastroenteritis

INTERVENTIONS:
Procedure: Stool sampling — Stool samples collected and checked for the presence of rotavirus
  Groups: Gastroenteritis cohort

SUMMARY:
The purpose of this study is to estimate the effectiveness of 2 doses of Rotarix™ vaccination in preventing rotavirus severe gastroenteritis among children hospitalized in Belem area, Brazil.

DETAILED DESCRIPTION:
The study will be comprised of two parts: Case-control study and Rotavirus strain surveillance.

ELIGIBILITY:
Inclusion Criteria:

For cases:

* A male or female child born after 6 March 2006 and at least 12 weeks of age.
* Subject admitted to the study clinics/hospitals for severe gastroenteritis during the study period.
* Onset of severe gastroenteritis ≤ 14 days prior to admission.
* Laboratory confirmed rotavirus positive stool sample at hospital admission or during the first 48 hours of hospitalization.
* Written informed consent obtained from the parent or guardian of the subject.

For controls:

* Admitted for non-gastroenteritis causes at the same clinic/hospital as the case.
* Living in the same neighbourhood as the case for at least three consecutive months without any symptoms of gastroenteritis or severe gastroenteritis on the day of interview of his/ her parents/ guardians.
* Being born within +- 2 weeks from the date of birth of the case. If the number required is not available, then the range would be extended to +- 4 weeks, and ultimately up to +- 6 weeks for hospital controls. For neighbourhood controls, the range may be extended to +- 8 weeks.
* Written informed consent obtained from the parent or guardian of the child.

Exclusion Criteria:

For cases:

* Subject has previously participated as case or control in this study.
* Onset of severe gastroenteritis > 48 hours after admission to the hospital (nosocomial infections).

For controls:

* For hospital controls: Child who has symptoms of gastroenteritis during current hospitalization or on the day of interview of his/her parent or guardian or for neighbourhood controls: Child who has symptoms of gastroenteritis or severe gastroenteritis on the day of interview of his/her parent or guardian.
* Exclude children with the following vaccine preventable diseases: measles, mumps, rubella, diphtheria, pertussis, tetanus, tuberculosis, invasive Haemophilus influenzae type B (Hib) infections (meningitis, bacteraemia, septic arthritis, cellulitis, and epiglottitis) and hepatitis B.
* Child has participated in the past as a case or control in this study.
* Child living in the same house as the case

Min Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastroenteritis Cohort: Cases will include children born after 6 March 2006, at least 12 weeks of age and hospitalized for rotavirus severe gastroenteritis the study clinics/hospitals, during the designated study period, Hospital control cohort: Children hospitalized for non gastroenteritis causes, Neighbourhood control cohort: Children without any symptoms of gastroenteritis or severe gastroenteritis.
Sampling Method: Non-Probability Sample
Enrollment: 1944 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Risk of Enzyme Linked Immunosorbent Assay (ELISA) confirmed rotavirus severe gastroenteritis in children fully vaccinated with Rotarix™, compared to risk of ELISA confirmed rotavirus severe gastroenteritis in unvaccinated children | Average time frame: 12-24 months

SECONDARY OUTCOMES:
Risk of ELISA confirmed rotavirus severe gastroenteritis in children vaccinated with at least one dose of Rotarix™, compared to risk of ELISA confirmed rotavirus severe gastroenteritis in unvaccinated children | Average time frame: 12-24 months
Occurrence of severe gastroenteritis among children admitted to study clinics/hospitals for severe gastroenteritis | Average time frame: 12-24 months
Occurrence of rotavirus serotypes among children | Average time frame: 36 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Belém, Pará, Brazil

REFERENCES:
- [Background] Justino MC, Linhares AC, Lanzieri TM, Miranda Y, Mascarenhas JD, Abreu E, Guerra SF, Oliveira AS, da Silva VB, Sanchez N, Meyer N, Shafi F, Ortega-Barria E, Soriano-Gabarro M, Colindres RE. Effectiveness of the monovalent G1P[8] human rotavirus vaccine against hospitalization for severe G2P[4] rotavirus gastroenteritis in Belem, Brazil. Pediatr Infect Dis J. 2011 May;30(5):396-401. doi: 10.1097/INF.0b013e3182055cc2. PMID 21150692